CLINICAL TRIAL: NCT01619345
Title: Pharmacoscintigraphic Investigation NN9924 in Healthy Male Subjects
Brief Title: Pharmacoscintigraphic Investigation of NN9924 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-3957; 2011-004162-14 (EudraCT Number); U1111-1123-7450 (Other: WHO)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1: NN9924 with 50 mL water (Experimental)
  Interventions: Drug: semaglutide
- Period 2: NN9924 with 240 mL water (Experimental)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Subjects will be treated with two single doses of 10 mg semaglutide in a tablet. Dosing will be done on 2 dosing visits separated by 4 to 6 weeks.
  Other Names: NN9924

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate whether the volume of water administered with NN9924 affects the anatomical location (stomach or proximal small bowel) of tablet erosion.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Body mass index (BMI) of 18.5-30.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Males who are not willing to use two acceptable forms of highly effective contraception
* Participation in another clinical trial within 90 days
* Any chronic disorder or severe disease
* Use of GLP-1 (glucagon-like peptide-1) agonists within 3 months preceding dosing
* Subjects who are smokers
* Subjects who have donated any blood or plasma in the past month or in excess of 500 mL within the 12 weeks preceding screening

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Anatomical location (stomach or proximal small bowel) of tablet at complete tablet erosion (CTE) | Assessed 0-4 hours post dose

SECONDARY OUTCOMES:
Area under the NN9924 concentration curve | From time 0-24 hours
Anatomical location of initial tablet erosion (ITE) | Assessed 0-4 hours post dose
Time to ITE | Assessed 0-4 hours post dose
Time to CTE | Assessed 0-4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Nottingham, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com